CLINICAL TRIAL: NCT02589145
Title: Lenalidomide Combined With Vorinostat/Gemcitabine/Busulfan/Melphalan With Autologous Stem-Cell Transplantation in Diffuse Large B-Cell Lymphoma of the ABC Subtype
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed due to very slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0558; NCI-2015-01938 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma
Keywords: Blood And Marrow Transplantation; Diffuse large B-cell lymphoma; DLBCL; Busulfan; Busulfex; Myleran; Lenalidomide; CC-5013; Revlimid; Vorinostat; SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza; Gemcitabine; Gemcitabine Hydrochloride; Gemzar; Melphalan; Alkeran; Rituximab; Rituxan; Dexamethasone; Decadron; Glutamine; Enterex; Glutapack-10; NutreStore; Resource; GlutaSolve; Sympt-X G.I.; Symptx-X; Pyridoxine; Enoxaparin; Lovenox Injection; Palifermin; Kepivance
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide; Vorinostat; Gemcitabine; Busulfan; Melphalan; Rituximab; Dexamethasone; Calcium Dobesilate; Glutamine; Health Resources; Pyridoxine; Enoxaparin; Stem Cell Transplantation; Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide + Vorinostat/Gem/Bu/Mel + AutoSCT (Experimental): Vorinostat and lenalidomide administered orally at the same time within 1 hour before the daily dose of chemotherapy.
  Gemcitabine administered as a loading dose of 75 mg/m2 followed by infusion on days -8 and -3.
  Busulfan test dose administered as outpatient before admission, or as inpatient on day -10. The "test dose" of 32 mg/m2 based on actual body weight. Doses of days -6 and -5 subsequently adjusted to target an AUC of 4,000 microMol.min-1.
  Melphalan administered at 60 mg/m2 on days -3 and -2.
  Patients with CD20+ tumors receive rituximab 375 mg/m2 on day -9 in the AM as an inpatient.
  Dexamethasone 8 mg by vein twice a day from day -8 to day -2. Caphosol oral rinses 30 mL four times a day used from day -8. Oral glutamine, 15 g four times a day, swished, gargled and swallowed started on day -8.
  Pyridoxine 100 mg by vein or mouth three times a day from day -1. Enoxaparin 40 mg subcutaneously daily from admission until platelet count drops below 50,000/mm3.
  Interventions: Drug: Lenalidomide; Drug: Vorinostat; Drug: Gemcitabine; Drug: Busulfan; Drug: Melphalan; Drug: Rituximab; Drug: Dexamethasone; Drug: Caphosol; Drug: Glutamine; Drug: Pyridoxine; Drug: Enoxaparin; Procedure: Stem Cell Transplant; Drug: Palifermin

INTERVENTIONS:
Drug: Lenalidomide — Dose Escalation Phase Starting dose of Lenalidomide: 50 mg by mouth on Days -9 to -2.
  Dose Expansion Phase Starting Dose: Maximum tolerated dose from Phase I.
  Other Names: CC-5013; Revlimid
Drug: Vorinostat — 1000 mg by mouth on Days -9 to -2.
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
Drug: Gemcitabine — Gemcitabine administered as a loading dose of 75 mg/m2 by vein on Day -8 and 2775 mg by vein on Day -3.
  Other Names: Gemcitabine Hydrochloride; Gemzar
Drug: Busulfan — Busulfan test dose administered by vein either as outpatient before admission, or as inpatient on day -10. The "test dose" of 32 mg/m2 based on actual body weight. Doses of days -6 and -5 subsequently adjusted to target an AUC of 4,000 microMol.min-1.
  Other Names: Busulfex; Myleran
Drug: Melphalan — 60 mg/m2 by vein on days -3 and -2.
  Other Names: Alkeran
Drug: Rituximab — Patients with CD20+ tumors receive Rituximab 375 mg/m2 by vein on day -9 in the AM as an inpatient.
  Other Names: Rituxan
Drug: Dexamethasone — 8 mg by vein twice a day from Day -8 AM to Day -2 PM.
  Other Names: Decadron
Drug: Caphosol — Caphosol oral rinses 30 mL four times a day used from Day -8.
Drug: Glutamine — Oral glutamine, 15 g four times a day, swished, gargled and swallowed started on Day -8.
  Other Names: Enterex; Glutapak-10; NutreStore; Resource; GlutaSolve; Sympt-X G.I.; Symptx-X
Drug: Pyridoxine — 100 mg by vein or mouth three times a day from Day -1
Drug: Enoxaparin — 40 mg subcutaneously daily from admission until platelet count drops below 50,000/mm3.
  Other Names: Lovenox Injection
Procedure: Stem Cell Transplant — Stem cell transplant performed on Day 0.
  Other Names: SCT
Drug: Palifermin — Palifermin per departmental standard of care with 3 doses to be administered prior to starting chemotherapy and 3 doses starting on day 0.
  Other Names: Kepivance

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of lenalidomide that can be given in combination with vorinostat, gemcitabine, busulfan, and melphalan, with a stem cell transplant, and with or without rituximab. Researchers also want to learn about the safety and effectiveness of this combination.

DETAILED DESCRIPTION:
Central Venous Catheter:

Many of the drugs given in this study and the stem cell transplant will be given by vein through a central venous catheter (CVC). A CVC is a sterile flexible tube and needle that will be placed into a large vein while you are under local anesthesia. Blood samples will also be drawn through your CVC. The CVC will remain in your body during treatment. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of lenalidomide based on when you join this study. Up to 3 dose levels of lenalidomide will be tested. At least 2 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of lenalidomide is found.

All participants will receive the same dose level of vorinostat, gemcitabine, busulfan, rituximab, and melphalan. However, if the first group of participants have any bad side effects, the dose level of gemcitabine may be lowered for all other groups.

Busulfan Test Dose:

In stem cell transplants, the days before you receive your stem cells are called minus days. The day you receive the stem cells is called Day 0. The days after you receive your stem cells are called plus days.

You will receive a test dose of busulfan by vein over about 60 minutes. This low-level test dose of busulfan is to check how the level of busulfan in your blood levels changes over time. This information will be used to decide the next dose needed to match your body size. You will most likely receive this as an outpatient during the week before you are admitted to the hospital. If it cannot be given as an outpatient, you will be admitted to the hospital on Day -11 (11 days before your stem cells are returned to your body) and the test dose will be given on Day -10.

Blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing of busulfan 11 times. PK testing measures the amount of study drug in the body at different time points and will help the study doctor determine what your dose of busulfan should be on study. These blood samples will be drawn at various timepoints before you receive busulfan and over about the next 11 hours. The blood samples will be repeated again on the first day of high-dose busulfan treatment (Day -8). A temporary heparin lock line will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for the PK tests to be performed, you will receive the standard fixed dose of busulfan.

You will also receive palifermin by vein over about 30 seconds each day to help decrease the risk of side effects in the mouth and throat either during the 2 days before you are admitted (inpatient) or during the 3 days before you are admitted (outpatient) You may ask the study staff about the risks of palifermin.

Study Drug Administration (all patients):

Beginning on Day -8, you will swish caphosol and glutamine liquids in your mouth 4 times a day, for about 2 minutes each time. You will swish these liquids every day until you leave the hospital. You will swallow the glutamine. These drugs are used to help decrease the risk of side effects in the mouth and throat.

On Days -9 through Day -2, you will take lenalidomide and vorinostat by mouth, with food.

If you the doctor thinks it is needed, you will receive rituximab by vein over 3-6 hours as part of standard of care, on Day -9.

On Day -8, you will receive gemcitabine by vein over 4½ hours.

On Days -8 through Day -5, you will receive busulfan by vein over 2 hours.

On Day -3, you will receive gemcitabine by vein over 4½ hours and then melphalan by vein over 30 minutes.

On Day -2, you will receive melphalan by vein over 30 minutes.

On Day -1, you will rest (you will not receive chemotherapy).

On Day 0, you will receive your stem cells by vein over about 30-60 minutes.

You will receive 3 more doses of palifermin by vein over 15-30 seconds on Days 0, +1, and +2.

As part of standard care, you will receive G-CSF (filgrastim) as an injection under your skin 1 time each day starting on Day +5 until your blood cell levels return to normal. You may ask the study staff about the risks of filgrastim.

Pregnancy Tests:

If you can become pregnant and have regular menstrual cycles, blood (up to 2 teaspoons) will be drawn for a pregnancy test on the following schedule:

* Within 10-14 days and within 24 hours before your first dose of lenalidomide, even if you have not had a menstrual period due to treatment or you have only had 1 menstrual period in the past 24 months.
* One (1) time each week for 4 weeks, then every 4 weeks while taking lenalidomide.
* Four (4) weeks after you stop taking lenalidomide.

If you have irregular menstrual cycles, you will have pregnancy tests every week for the first 28 days, then every 14 days while you are taking lenalidomide, again when you have been taken off of lenalidomide therapy, and then 14 and 28 days after you have stopped taking lenalidomide.

Length of Study:

As part of standard care, you will remain in the hospital for about 3-4 weeks after the transplant. After you are released from the hospital, you will continue as an outpatient in the Houston area to be monitored for infections and transplant-related complications.

You will be taken off study about 100 days after the transplant. You may be taken off study early if the disease gets worse, if intolerable side effects occur, if you are unable to follow study directions, or if you choose to leave the study early.

If for any reason you want to leave the study early, you must talk to the study doctor. It may be life-threatening to leave the study after you have started to receive the study drugs but before you receive the stem cell transplant because your blood cell counts will be dangerously low.

Follow-Up:

About 100 days after the transplant:

* You will have a physical exam.
* Blood (about 4 teaspoons) and urine will be collected for routine tests and to check your kidney and liver function.
* If the doctor thinks it is needed, you will have computed tomography (CT) and/or positron emission tomography (PET) scans to check the status of the disease.
* If the doctor thinks it is needed, you may have a bone marrow aspiration and biopsy to check the status of the disease. To collect a bone marrow aspiration/biopsy, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.

This is an investigational study. Lenalidomide is FDA approved and commercially available for the treatment of multiple myeloma (MM) and myelodysplastic syndrome (MDS). Rituximab is FDA approved and commercially available for the treatment of non-Hodgkin's lymphoma and certain types of leukemia. Vorinostat is FDA approved and commercially available for the treatment of cutaneous T-cell lymphoma (CTCL). Gemcitabine is FDA approved and commercially available for the treatment of non-small cell lung cancer (NSCLC), breast cancer, pancreatic cancer, and ovarian cancer. Busulfan is FDA approved and commercially available for the treatment of chronic myeloid leukemia (CML). Melphalan is FDA approved and commercially available for the treatment of lymphoma.

The use of these study drugs in combination to treat DLBCL is considered investigational. The study doctor can explain how the study drugs are designed to work.

Up to 30 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-65
2. Patients with ABC (determined by immunohistochemistry using the Hans algorithmI) DLBCL with primary refractory disease, relapse <12 months after initial therapy, secondary International Prognostic Index (IPI) >1, less than partial response to salvage treatment or exposure to >3 salvage regimens
3. Adequate renal function, as defined by an estimated serum creatinine clearance >/= 50 ml/min (MDRD method) and/or serum creatinine </= 1.8 mg/dL
4. Adequate hepatic function (SGOT and/or SGPT </= 3 x ULN; bilirubin and ALP </= 2 x ULN
5. Adequate pulmonary function with FEV1, FVC and DLCO (corrected for Hgb) >/= 50%
6. Adequate cardiac function with left ventricular ejection fraction >/= 40%. No uncontrolled arrhythmias or symptomatic cardiac disease
7. ECOG performance status <2
8. Negative Beta HCG in woman with child-bearing potential
9. All study participants must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of the REMS program.
10. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program.

Exclusion Criteria:

1. Grade >/= 3 non-hematologic toxicity from previous therapy that has not resolved to </= G1
2. Prior whole brain irradiation
3. Active hepatitis B, either active carrier (HBsAg +) or viremic (HBV DNA >/= 10,000 copies/mL, or >/= 2,000 IU/mL)
4. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology
5. Active infection requiring parenteral antibiotics
6. HIV infection, unless receiving effective antiretroviral therapy with undetectable viral load and normal CD4 counts
7. Radiation therapy in the month prior to enrollment
8. History of arterial thromboembolic events in the past 3 months and of venous thromboembolic events in the past month
9. History of hypersensitivity of lenalidomide or thalidomide

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled at MD Anderson Clinic starting on August 22, 2016.
Groups:
- Lenalidomide Dose Level 1: Lenalidomide 50 mg PO for 8 days+Vorinostat 1000 mg PO for 8 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto Stem Cell Transplant (SCT)
- Lenalidomide Dose Level 2: Lenalidomide 75 mg PO for 8 days+Vorinostat 1000 mg PO for 8 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto Stem Cell Transplant (SCT)
- Lenalidomide Dose Level 3: Lenalidomide 100 mg PO for 8 days+Vorinostat 1000 mg PO for 8 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto Stem Cell Transplant (SCT)
Period: Overall Study
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
Started | 4 | 2 | 2
Completed | 4 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients age 15-65 with ABC (determined by immunohistochemistry using the Hans algorithm) Diffuse Large B-cell Lymphoma (DLBCL) with primary refractory disease.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3 | Total
Number analyzed (Participants) | 4 | 2 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 2 | 8
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 55.5 [36 to 59] | 42.5 [21 to 64] | 58 [54 to 62] | 56.5 [21 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 3 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 2 | 8
Disease Status [Count of Participants; unit: Participants] — Disease Status at time of Transplant (Complete remission, Partial Remission, Stable Disease, or Progressive Disease) Population: Patients age 15-65 with ABC (determined by immunohistochemistry using the Hans algorithm) Diffuse Large B-cell Lymphoma (DLBCL) with primary refractory disease..
  Participants
    Complete Remission | 3 | 2 | 1 | 6
    Partial Remission: number analyzed (Participants) | 1 | 0 | 1 | 2
    Partial Remission | 1 |  | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Established the maximum tolerated dose (MTD) of lenalidomide combined with vorinostat/gemcitabine/busulfan/melphalan with autologous stem-cell transplant ASCT). Maximum tolerated dose (MTD) of lenalidomide based on DLT was defined as any Grade 4 or 5 nonhematologic, noninfectious toxicity or any grade 3 mucositis or skin toxicity lasting > 5 days at their peak severity. Lenalidomide doses were chosen adaptively for successive cohorts with a minimum size of 2 patients. Toxicity scoring followed the National Cancer Institute Common Toxicity Criteria, version 4.
Time Frame: Enrollment up to day 30 post transplant for each dosing cohort
Population: Due to low accrual, MTD could not be determined for this outcome.
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Event-free Survival (EFS)
Description: Determined the 2-year event-free survival (EFS)
Time Frame: Up to 2 years post transplant
Population: Due to low accrual, EFS could not be determined for this outcome.
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Assessed the 2-year overall survival (OS)
Time Frame: Up to 2 years post transplant
Population: Due to low accrual, OS could not be determined for this outcome.
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Complete Remission (CR) Rate
Description: Determined complete remission (CR) rate
Time Frame: Up to 2 years post transplant
Population: Due to low accrual, CR rate could not be determined for this outcome.
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Overall Remission Rate (ORR)
Description: Determined overall remission rate (ORR) rate
Time Frame: Up to 2 years post transplant
Population: Due to low accrual, the ORR could not be determined for this outcome.
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Toxicity Profile
Description: Determined the toxicity profile
Time Frame: Up to 2 years post transplant
Population: Due to low accrual, the Toxicity profile could not be determined for this outcome.
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Pharmacodynamic Studies
Description: Evaluated IRF4, SPIB, STAT1, p-STAT1, CARD11, I-kappa-Kinase-beta and p-I-kappa-Kinase-beta in PBMNC pre- and post-treatment (at baseline and on day -1).
Time Frame: Up to 2 years post transplant
Population: Due to low accrual, the pharmacodynamic studies could not be determined for this outcome.
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 100 Days post autologous transplant
Arm/Group | Lenalidomide Dose Level 1 | Lenalidomide Dose Level 2 | Lenalidomide Dose Level 3
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Dose Level 1 (N=4) | Lenalidomide Dose Level 2 (N=2) | Lenalidomide Dose Level 3 (N=2)
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis (Gastrointestinal disorders) | 1 | 0 | 0
Elevated Bilirubin (Hepatobiliary disorders) | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide Dose Level 1 (N=4) | Lenalidomide Dose Level 2 (N=2) | Lenalidomide Dose Level 3 (N=2)
Fluid Overload (General disorders) | 3 (3) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Neutropenic Fever (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Transaminitis (Hepatobiliary disorders) | 2 (2) | 2 (3) | 1 (2)
Elevated Bilirubin (Hepatobiliary disorders) | 4 (4) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Skin other Desquamation/Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (2) | 1 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT02589145/Prot_SAP_000.pdf